CLINICAL TRIAL: NCT03129074
Title: A Phase 2, Single Arm Study of Varlitinib Plus Capecitabine in Patients With Advanced or Metastatic Biliary Tract Cancer as First-line Systemic Therapy
Brief Title: Study of Varlitinib Plus Capecitabine in Patients With Advanced or Metastatic Biliary Tract Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-016
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Advanced or Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Varlitinib given in combination with capecitabine (Experimental): * PO varlitinib 300 mg BID
  * PO capecitabine 1000 mg/m2 BID
  Interventions: Drug: Varlitinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Varlitinib — everyday
Drug: Capecitabine — from Day 1 to Day 14 followed by 7-day of rest period, every 21 days.

SUMMARY:
The purpose of the study is to assess the efficacy of varlitinib in combination with capecitabine as measured by objective response rate (ORR) assessed by independent central review (ICR), based on RECIST v1.1 criteria.

DETAILED DESCRIPTION:
Also to explore the role of biomarkers as predictors of response and clinical benefit with varlitinib

ELIGIBILITY:
Inclusion Criteria:

1. Are of or older than the legal age in the respective countries at the time when written informed consent is obtained.
2. Are able to understand and willing to sign the informed consent form.
3. Have histologically confirmed diagnoses of relapsed, locally advanced (unresectable) or metastatic biliary tract cancer, including intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer and carcinoma of Ampulla of Vater.
4. Have eligible tumor tissue (archival or fresh) for the evaluation of relevant primary endpoints.

   (Note: For patients without eligible tumor tissue, a discussion with the sponsor is mandatory).
5. Have radiographically measurable disease as determined by the investigator based on the RECIST v1.1 criteria.
6. Have no evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below 1.5 x upper level of normal (ULN).
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Have an estimated life expectancy of more than 3 months, at the time of screening.
9. Have adequate organ and hematological function:

   1. Hematological function, as follows:

      * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
      * Platelet count ≥ 100 x 109/L
   2. Renal functions, as follows:

      * estimated glomerular filtration rate (eGFR) or creatinine clearance (CrCl) > 50 mL/min/1.73m2
   3. Hepatic function, as follows:

      * Total bilirubin ≤ 1.5 x ULN
      * aspartate aminotransferase and alanine aminotransferase ≤ 5 x ULN

Exclusion Criteria:

1. Have received systemic anti-cancer treatment except (neo-) adjuvant therapy for early stage disease.
2. Are currently on or have received radiation or local treatment within the past 4 weeks for the target lesion(s), prior to screening.
3. Had undergone major surgical procedures within 28 days prior to study cycle 1 day 1.
4. Have a metastatic brain lesion(s), including asymptomatic and well controlled lesion(s).
5. Have malabsorption syndrome, diseases significantly affecting gastrointestinal function, or difficulty in swallowing and retaining oral medications.
6. Have any history of other malignancy unless in remission for more than 1 year (skin carcinoma and carcinoma-in-site of uterine cervix treated with curative intent is not exclusionary).
7. Are female patients who are pregnant or breast feeding.
8. Have been previously treated with varlitinib or capecitabine.
9. Have received any investigational drug (or have used an investigational device) within the last 14 days before receiving the first dose of study medication.
10. Have unresolved or unstable serious toxicity (≥ CTCAE 4.03 Grade 2), with the exception of anemia, asthenia, and alopecia, from prior administration of another investigational drug and/or prior anti-cancer treatment.
11. Have a known positive test for human immunodeficiency virus, active viral hepatitis C, viral hepatitis B infection with hepatitis B virus DNA exceeding 2000 IU/mL.
12. Have a known history of drug addiction within last 1 year, on the basis of which there could be a higher risk of non-compliance to study treatment.
13. Need continuous treatment with proton pump inhibitors during the study period.
14. Have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis, or with a history of interstitial lung disease or current interstitial lung disease.
15. Have any history or presence of clinically significant condition which in the opinion of the investigator could jeopardize the safety of the patient or the validity of the study results.
16. Have a baseline corrected QT interval > 450 ms or patients with known long QT syndrome, torsade de pointes, symptomatic ventricular tachycardia, unstable cardiac syndrome in the past 3 months before screening visit, > class 2 NYHA (The New York Heart Association Functional Classification heart failure), > grade 2 CCS (the Canadian Cardiovascular Society Guidelines) angina pectoris, or receiving quinidine, procainamide, disopyramide, amiodarone, dronedarone, arsenic, dofetilide, or sotalol methadone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Are of or older than the legal age in the respective countries at the time when written informed consent is obtained.
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study duration, estimated 3 years
  Number (%) of patients with at least one visit response of CR or PR. Tumor evaluations will continue until the earlier of disease progression or starting a subsequent anti-cancer therapy.
Biomarker | Through study duration, estimated 3 years
  Use Next generation sequencing/Immunohistochemistry to identify relationships between response to varlitinib and mutations or overexpression in human epidermal growth factor receptor (HER) receptors and the downstream signaling proteins, as well as, mutations in selected cancer pathways.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study duration, estimated 3 years
  Defined as the time from start of treatment until the date of objective disease progression or death (by any cause in the absence of disease progression).
Overall survival (OS) | Through study duration, estimated 3 years
  Defined as the time from start of treatment until death by any cause.
Duration of response (DoR) | Through study duration, estimated 3 years
  Defined as the time, in days, from the first recorded achievement of a response (PR or above) until time of objective disease progression in the subset of patients classified as responders in the assessment of ORR
Disease control rate (DCR) | Through study duration, estimated 3 years
  Defined as the proportion of patients with a best response of stable disease maintained for at least 12 weeks (-5 days), PR or CR as defined by RECIST v1.1 criteria.
Objective response rate (ORR) | Through study duration, estimated 3 years
  Defined as the proportion of patients with a best objective response (BOR) of complete response (CR) or partial response (PR), as assessed by the investigator defined by the RECIST v1.1 criteria.
Incidence of Adverse Events and changes from baseline in safety parameters | Through study duration, estimated 3 years
  Incidence of Adverse Events, categorized in accordance to CTCAE 4.03 and changes from baseline in safety parameters (including vital signs, ECG parameters, clinical laboratory tests).

IPD SHARING:
Plan to Share IPD: No